CLINICAL TRIAL: NCT00985309
Title: Clinical Parameters Predicting Unsatisfactory Cervicovaginal Cytology in Conventional Smears
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Chien-Hsing Lu, Department of OB/GYN, Taichung Veterans General Hospital
Other Study IDs: C08213
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Unsatisfactory Pap Smear
Keywords: unsatisfactory; Pap smear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
According the terminology of Bethesda 2001, the unsatisfactory cervical cytology can be categorized into specimen rejected, or specimen processed and examined, but unsatisfactory for evaluation of epithelial abnormality. Most of the unsatisfactory cervical cytology was due to scanty epithelial cells, which was defined by less than an estimated 8,000 to 12,000 well-visualized squamous cells for conventional smears. Follow-up of unsatisfactory smear found an increased rate of cervical preinvasive and invasive lesions. Thus, an unsatisfactory smear deserves careful follow-up and studies. Although the Bethesda system allows criteria modification in cases of hysterectomy, pelvic irradiation therapy, or chemotherapy, no studies investigated the clinical factors related to the incidence of unsatisfactory smear. Thus, the investigators designed this trial to study the clinical factors relating to unsatisfactory cervicovaginal smear.The list of patients who received Papanicolaou smear between March 2006 and August 2006 in our hospital will be obtained from the Pathological Department first. Then the investigators will review the medical records from HIS system and pathologic files of these patients. On estimation, 7,437 cases will be enrolled for analysis. Clinical parameters for analysis include: age, gravidity, parity, abortion, menopause, location of Pap smear, history of pelvic malignancy, pelvic irradiation, cervical conization, hysterectomy; at pregnancy; three months postpartum; vaginal bleeding, vaginal abnormal discharge, intrauterine device, and cervical polyp found during pelvic examinations. Patients who missed any of above data will be excluded for analysis. The investigators will use univariate and multivariate analysis for data processing and statistic analysis to find out the relationship between clinical parameters and unsatisfactory cervicovaginal Pap smears.

ELIGIBILITY:
Inclusion Criteria:

* A cohort of consecutive patients who received conventional Pap smear between March 2006 and August 2006 in Taichung Veterans General Hospital

Exclusion Criteria:

* nil

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of consecutive patients who received conventional Pap smear between March 2006 and August 2006 in Taichung Veterans General Hospital
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
unsatisfactory Pap smear rates in various clinical conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of OB/GYN, Taichung Veterans General Hospital, Taichung, Taiwan